CLINICAL TRIAL: NCT02608255
Title: A Prospective Pilot Study to Evaluate a New Marker of Ischemia in Chest Pain Triage
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2015-A01378-41
Record Dates: First submitted 2015-11-10; First posted 2015-11-18 (Estimated); Last update posted 2017-01-04 (Estimated); Status verified 2017-01

CONDITIONS: Acute Coronary Syndrome
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- acute coronary syndromes (Experimental)
  Interventions: Other: blood samples

INTERVENTIONS:
Other: blood samples

SUMMARY:
A Single-center prospective pilot study enrolling chest pain patients. CD 26 measurement will be performed and compared to troponin µs for early triage of these patients. This novel biomarker of myocardial ischemia (CD26) will be measured at the time of first medical contact (T0) and after 30 min simultaneously o troponin Ic.

All patients aged over 18 years with chest pain which may be related to acute coronary syndrome requiring pre hospital medical contact through the Emergency Medical Service.

DETAILED DESCRIPTION:
First objectives: demonstrating the early positivity of CD26 compared to ultra-sensitive troponin.

ELIGIBILITY:
Inclusion Criteria:

* Subject with compatible symptoms with an acute coronary syndrome, for at least 15 minutes and not older than 3 hours (eg discomfort, tightness or chest pain, pain radiating to the left arm or two arms, pain in the jaw, pain in the back / neck / stomach, breathlessness , cold sweats, nausea / vomiting , dizziness )
* Man or woman,
* Patient Did not receive heparin or low molecular weight heparin (LMWH ) before the initial blood sample ,
* Patient Agreeing to participate in the study and who signed an informed consent

Exclusion Criteria:

* Minor or major patient trust
* Patient Not having signed informed consent (refusal , physical or mental disability ... )
* Patient Who received anticoagulation before carrying blood samples
* Patient With a progressive septic processes , neoplasia undergoing treatment, dialyzed kidney failure, a history of surgery or coronary angioplasty less than six months.
* Transplanted heart, renal or hepatic
* heart attack
* Subject Whose symptoms clearly eliminates acute coronary syndrome ( penetrating trauma, traumatic injury by crushing ... )
* Patient Died between the time of inclusion and arrival in the cardiology intensive care ( SIC )
* Patient Withdrawing consent under study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2016-01; Primary Completion 2016-11 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
blood sample : dosage of CD26 | 12 MONTHS
  demonstrating the early positivity of CD26 compared to ultra-sensitive troponin.
blood sample: dosage of the copeptin | 12 months
blood sample: dosage of troponin | 12 months
blood sample : dosage of IMA | 12 months
  IMA (Albumin modified by the ischaemia)
blood sample: dosage of adenosin | 12months

CONTACTS AND LOCATIONS:
Overall Officials: BONELLO laurent, Principal Investigator — AP HM
Locations (1):
- Assistance Publique Hopitaux de Marseille, Marseille, France